CLINICAL TRIAL: NCT02408497
Title: Evaluation of the Use of Non-invasive 4D Ultrasound Clarity System in Real-time Tracking of the Target Volume in Prostate IMRT/RapidArc Therapy
Brief Title: Use of Non-invasive 4D Ultrasound Clarity System in Prostate IMRT/RapidArc Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: NCC DRO 4D-us CS
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A single arm phase II study of prostate motion for prostate cancer to primarily compare prostate motion between different treatment duration for IMRT and VMAT.

DETAILED DESCRIPTION:
Primarily, this is a single arm phase I study of prostate motion for prostate cancer to primarily compare prostate motion between different treatment duration for IMRT and VMAT. The radiation therapy is to be delivered using intensity modulated radiotherapy (IMRT) or Volumetric Modulated Arc therapy (VMAT) with the aid of volumetric image guidance to ensure accuracy and real-time 3D ultrasound images as observational record of the prostate motion. All the recruited patients are prescribed and treated with either VMAT or IMRT treatment. In order to simulate the behaviour of prostate motion in an IMRT scenario, the group of VMAT patients will be required to remain in treatment position for an additional 7 minutes depending on techniques used (once a week).

In order to assess the level of acceptance of the treatment position, responses to the same comfort survey for the current treatment position (i.e. using leg immobiliser) by a cohort of 60 patients treated in another IGRT treatment room will be used as the baseline. In addition, RTT satisfaction questionnaire will also be administered to assess the handling of the new immobilizer.

Acute toxicity will be measured at preset intervals using CTCAE version 3.0 and as will International prostate symptom score (IPSS) questionnaire which focuses on urinary symptoms. Symptoms or toxicities reported from this study is relevant for patients treated with IMRT or VMAT with full bladder protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* Patient who cannot abide to the departmental hydration protocol
* Prostatectomy cases
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatment involved in this protocol requires contact of ultrasound probe to the perineum area.
* Patient enrolled in other clinical trials

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients who are going to receive IMRT/RapidArc therapy at site and are not participating any other clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The extent of intra-fraction prostate motion using an ultrasound system during IMRT and during RapidArc therapy | 2 years

SECONDARY OUTCOMES:
The 3D ultrasound capability of the Clarity® system (from Elekta AB Stockholm, Sweden) in providing real-time information of the prostate movement during the treatment delivery | 2 years
The efficacy of full bladder protocol for patient undergoing prostate radiotherapy | 2 years
The rate of acute GI and GU side effects within 3 months (<90 days) after radical radiotherapy | 2 years
Patient comfort, compliance and tolerance of two setup techniques | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kit Long Tuan, Dr, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore